CLINICAL TRIAL: NCT03092141
Title: Physical Training in Patients With Relapsing Polychondritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Samuel Katsuyuki Shinjo, PhD, Principal Investigator, University of Sao Paulo
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MYO-HCFMUSP-04
Record Dates: First submitted 2017-03-10; First posted 2017-03-27 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Physical Activity
MeSH Terms: conditions — Motor Activity | interventions — Physical Conditioning, Human; Exercise

STUDY DESIGN:
Intervention Model Description: Patients will submitted to physical training (12-weeks, twice/week)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients (Active Comparator): Patients will be submitted to physical training (12-weeks, twice/week)
  Interventions: Other: Physical training
- Control group (Active Comparator): Healthy individuals will be submitted to physical training (12-weeks, twice/week)
  Interventions: Other: Physical training

INTERVENTIONS:
Other: Physical training
  Other Names: Exercises

SUMMARY:
Physical training may improve physical capacity and health parameters in various systemic autoimmune diseases. Therefore, the present study will assess the role of an exercise training program in patients with relapsing polychondritis.

DETAILED DESCRIPTION:
Impact of physical training in patients with relapsing polychondritis.

ELIGIBILITY:
Inclusion Criteria:

* Fullfill the classification criteria of McADAM et al. (1976)
* Using prednisone ≤ 0.5 mg/kg/day in the last three months
* Sedentary

Exclusion Criteria:

* Disease relapsing
* Overlapping disease
* Chronic and/or current infections (viral, bacterial or fungal)
* Patients undergoing major surgery within six months before the study
* With commitment to ambulation (joint affection in limbs)
* Smoking
* Diabetes mellitus

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2021-04-29 (Actual); Study Completion 2021-04-29 (Actual)

PRIMARY OUTCOMES:
Cardiopulmonary test | 12 weeks
  Patients will undertake a maximal graded exercise test on a treadmill, with increments in velocity and grade at every minute until volitional exhaustion. VO2peak will be considered as the average of the final 30 s of the test. Ventilatory threshold (VAT) will be determined when ventilatory equivalent for VO2 (VE/VO2) increased without a concomitant increase in ventilatory equivalent for carbon dioxide (VE/VCO2). Respiratory compensation point (RCP) will be determined when VE/VO2 and VE/VCO2 increased simultaneously.

SECONDARY OUTCOMES:
Strength muscle tests | 12 weeks
  The dynamic 1-RM for the leg-press and the bench-press exercises, arm curl (with the dominant arm), and isometric strength (assessed by handgrip, with the dominant arm) will be assessed at baseline and after the intervention.
Healthy Assessment Questionnaire (HAQ) | 12 weeks
  Especific questionnaire to assess the quality of life. Pontuaction: 0.00-3.00
Functional muscle tests | 12 weeks
  Muscle function will be evaluated through the TUG and the TST tests
Muscle biopsy | 12 weeks
  After local anesthesia, a cutaneous incision will be made in lateral thigh face. The biopsy will be done using the Bergstrom needle. Histological (hematoxylin and eosin)/immunohistochemical (CD4, CD8, CD68, CD20, C5b-9, MHCI, MHCII, CD31) analysis will be performed in muscle samples (at baseline and after 12 weeks) in all patients (present study)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel K Shinjo, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- Samuel Katsuyuki Shinjo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No